CLINICAL TRIAL: NCT03045497
Title: Contrast-Enhanced Ultrasound for the Evaluation of Transarterial Chemoembolization With Drug Eluting Beads
Brief Title: Contrast-Enhanced Ultrasound in Predicting Treatment Response in Patients With Liver Cancer Receiving Transarterial Chemoembolization With Drug Eluting Beads
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12D.614; JT 2999 (Other: JeffTrial Number)
Record Dates: First submitted 2017-01-31; First posted 2017-02-07 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — perflutren; Dynamic Contrast Enhanced Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (contrast-enhanced ultrasound) (Experimental): Patients receive perflutren lipid microspheres IV and then undergo contrast-enhanced ultrasound imaging over approximately 1 hour prior to transarterial chemoembolization with drug eluting beads, at 1-2 weeks and 1 month post transarterial chemoembolization with drug eluting beads. Patients also undergo contrast-enhanced MRI at 1 month post-treatment per standard of care.
  Interventions: Drug: Perflutren Lipid Microspheres; Device: Dynamic Contrast-Enhanced Ultrasound Imaging; Device: Contrast-enhanced Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Perflutren Lipid Microspheres — Given IV
  Other Names: Definity
Device: Dynamic Contrast-Enhanced Ultrasound Imaging — Undergo contrast-enhanced ultrasound imaging
Device: Contrast-enhanced Magnetic Resonance Imaging — Undergo contrast-enhanced Magnetic Resonance Imaging
  Other Names: Contrast-enhanced MRI

SUMMARY:
This pilot clinical trial compares the use of contrast-enhanced ultrasound to contrast-enhanced magnetic response imaging (MRI), the current clinical standard, in predicting treatment response in patients with liver cancer receiving transarterial chemoembolization with drug eluting beads. Comparing results of diagnostic procedures before and after transarterial chemoembolization may help doctors predict a patient's response to treatment and help plan the best treatment. It is not yet known if contrast-enhanced ultrasound works better than contrast-enhanced MRI in predicting treatment response in patients with liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate if contrast-enhanced ultrasound of hepatocellular carcinomas at one to two weeks and one month correlate with the clinical evaluation standard of a contrast-enhanced MRI at one month (the current clinical standard) in patients who have undergone transarterial chemoembolization with drug eluting beads.

SECONDARY OBJECTIVES:

I. Establish whether changes in quantitative blood flow parameters relative to baseline correlate with effective embolization.

ELIGIBILITY:
Inclusion Criteria:

* Be scheduled for a transarterial chemoembolization using drug eluting beads for treatment of hepatocellular carcinoma
* Be medically stable
* If a female of child-bearing potential, must have a negative pregnancy test
* Have signed Informed Consent to participate in the study

Exclusion Criteria:

* Females who are pregnant or nursing
* Patients who are medically unstable, patients who are seriously or terminally ill, and patients whose clinical course is unpredictable; for example:

  * Patients on life support or in a critical care unit
  * Patients with unstable occlusive disease (eg, crescendo angina)
  * Patients with clinically unstable cardiac arrhythmias, such as recurrent ventricular tachycardia
  * Patients with uncontrolled congestive heart failure (New York Heart Association [NYHA] class IV)
* Patients with recent cerebral hemorrhage
* Patients with clinically significant and unstable renal disease (eg, transplant recipients in rejection)
* Patients who have undergone surgery within 24 hours prior to the study sonographic examination
* Patients with known hypersensitivity to perflutren
* Patients who have received any contrast medium (x-ray, MRI, computed tomography [CT], or ultrasound [US]) in the 24 hours prior to the research US exam
* Patients with cardiac shunts
* Patients with congenital heart defects
* Patients with severe emphysema, pulmonary vasculitis, or a history of pulmonary emboli
* Patients with respiratory distress syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-12-12 (Actual); Primary Completion 2013-12-05 (Actual); Study Completion 2013-12-05 (Actual)

PRIMARY OUTCOMES:
Ability of contrast-enhanced ultrasound to predict response to transarterial chemoembolization with drug eluting beads | Up to 1 month after transarterial chemoembolization
  Contrast-enhanced ultrasound of hepatocellular carcinomas at one month will be evaluated to see if it correlates with the clinical evaluation standard of a contrast-enhanced MRI at one month. Sensitivity, specificity, accuracy, positive predictive value, and negative predictive value will be calculated for the contrast-enhanced ultrasound exam. Correlations between these findings and both contrast-enhanced MRI findings and patient outcomes will be compared using the Fisher exact test. Inter- and intra-observer variability will also be calculated.

SECONDARY OUTCOMES:
Change in quantitative blood flow parameters | Baseline to up to 1 month after transarterial chemoembolization
  Whether changes in quantitative blood flow parameters relative to baseline correlate with effective embolization will be established.
Quantitative parameters of tumor vascularity | Baseline to up to 1 month after transarterial chemoembolization
Changes in perfusion | Baseline to up to 1 month after transarterial chemoembolization
Changes in contrast fill time | Baseline to up to 1 month after transarterial chemoembolization

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Forsberg, PhD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University

REFERENCES:
- See also: Sidney Kimmel Cancer Center — http://www.kimmelcancercenter.org
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/